CLINICAL TRIAL: NCT00417638
Title: A Randomized, Controlled Study of the Use of Central Venous Catheter Core Cooling Combined With Cold Saline, and Rewarming as an Adjunct to Percutaneous Coronary Intervention For the Treatment of Acute Myocardial Infarction
Brief Title: Rapid Intravascular Cooling in Myocardial Infarction as Adjunctive to Percutaneous Coronary Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZOLL Circulation, Inc., USA (Industry)
Collaborators: Lund University Hospital (Other); Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rapid MI-ICE-Pilot
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2010-01

CONDITIONS: Acute Anterior Myocardial Infarction
Keywords: myocardial infarction; acute intervention; percutaneous intervention; endovascular cooling; endovascular rewarming
MeSH Terms: conditions — Anterior Wall Myocardial Infarction; Myocardial Infarction | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients with acute STEMI - treatment with Hypothermia +PCI (Experimental): Hypothermia using endovascular cooling with the Celsius Control System as an adjunct therapy.
  Hypothermia before reperfusion by a combination of infusion of cold saline and endovascular catheter cooling as an adjunct therapy in patients with a STEMI scheduled to undergo primary percutaneous coronary intervention (PCI).
  Interventions: Device: Endovascular cooling by the Celsius Control System
- Patients with an acute STEMI eligible for primary PCI (Active Comparator): Standard of care treatment or the control group Patients with an acute STEMI eligible for primary PCI
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: Endovascular cooling by the Celsius Control System
  Arms: patients with acute STEMI - treatment with Hypothermia +PCI
Other: Standard of care
  Arms: Patients with an acute STEMI eligible for primary PCI

SUMMARY:
Rapid MI-ICE-Pilot is designed to demonstrate the safety and efficacy of the Celsius Control™ System (CCS) endovascular catheter to reduce the infarct size resulting from acute anterior myocardial infarction when used in combination with cold saline as an adjunct to immediate percutaneous coronary intervention (PCI) in patients with an occluded infarct-related artery.

DETAILED DESCRIPTION:
The CCS is an endovascular thermal control system that circulates cooled saline through an indwelling central venous catheter in a closed-loop manner. The system has received 510(k) approval from the FDA for use in temperature management in neuro-surgical and cardiac patients during surgery and in recovery/intensive care. It has also received European CE mark and Australian TGA approval. Animal data in a model of acute myocardial infraction support the hypothesis that rapid cooling, prior to acute PCI, may reduce infarct size. Meta-analysis of the previous acute MI trials ICE-IT (N = 228; 1:1 randomization, hypothermia : control, Innercool Therapies, Inc.) and COOL MI-I (Radiant Medical, Inc) suggests there is a reduction in infarct size as measured by 30-day SPECT in the population of patients with anterior MIs who were cooled below 35 C prior to PCI.

This study is designed to investigate the safety, feasibility and efficacy of rapid endovascular cooling in the setting of acute PCI in patients with anterior infarctions.

ELIGIBILITY:
Inclusion Criteria:

Each eligible patient must meet the following inclusion criteria :

1. Have ECG evidence of ongoing acute anterior myocardial infarction, involving a large area of myocardium, as defined by the following ECG criteria: a. Anterior infarct: ST-segment elevation >0.2mV measured 0.08 sec after the J point in 2 or more anatomically contiguous precordial leads, V1 through V4; and/or >0.2mV in lead V5 V6
2. Present to the RAPID MI-ICE site within six (6) hours of the onset of acute cardiac ischemic signs or symptoms (such as chest pain or pressure, arm or jaw pain, dyspnea, nausea/vomiting, or syncope)
3. Be a candidate for PCI and have PCI planned as the immediate intervention.
4. Be willing and able to comply with study procedures, including returning for the MRI scan at 4 ±2 days and return for the clinical examination on Day 30
5. Provide written informed consent prior to the initiation of study-specific procedures
6. Be in Killips Class I

Exclusion Criteria:

Patients are not eligible for the study if they meet one or more of the following criteria:

1. Age less than eighteen (<18) years of age
2. Age greater than seventy-five (>75) years of age
3. Are pregnant
4. Have a suspected aortic dissection
5. History of a prior anterior myocardial infarct or prior large myocardial infarct.
6. The suspected etiology of myocardial infarction is primarily related to substance abuse (e.g., cocaine, methamphetamine, etc.)
7. Acute administration of a thrombolytic agent for the qualifying MI
8. If (during the screening process) the determination is made by site-study personnel that initiation of cooling prior to diagnostic coronary angiography is technically not feasible for any reason (should the patient be randomized to the Hypothermia Arm), the prospective subject should not be enrolled
9. Require an immediate surgical or procedural intervention other than PCI (e.g. CABG)
10. Present in cardiogenic shock or with end-stage cardiomyopathy
11. Have undergone at least ten (10) minutes of cardiopulmonary resuscitation (CPR) prior to presentation to the PCI facility
12. History of previous MI with known, pre-existing, anterior pathologic Q-waves
13. History of surgical coronary artery revascularization (e.g., CABG, MIDCAB, or OPCAB)
14. Recent stroke (within 3 months)
15. Active bleeding, coagulopathy, or other contraindication to the placement of a heparin-coated 14F central venous catheter via a 14F femoral venous introducer sheath (e.g., known history of heparin induced thrombocytopenia, or IVC filter)
16. Contraindications to hypothermia, such as patients with known hematologic dyscrasias which affect thrombosis (e.g., cryoglobulinemia, sickle cell disease, serum cold agglutinins) or vasospastic disorders (such as Raynaud's or thromboangitis obliterans)
17. Personal or familial history of malignant hyperthermia
18. Known end-stage renal disease (ESRD; e.g., on dialysis, or status-post renal transplant), known hepatic failure (e.g., cirrhosis, or acute hepatitis), or any other contraindication to receiving meperidine (such as use of MAO inhibitors within previous 14 days, history of seizures, history of hypersensitivity to meperidine, etc.) [Note: Patients with a contraindication to buspirone administration may be enrolled but should not be given buspirone as part of the anti-shivering regimen.]
19. Any other acute or chronic condition which the Investigator believes will unacceptably increase the risk of study participation or interfere with study procedures and assessments
20. Deemed unsuitable by the investigators to participate in the study.
21. Signs of cardiogenic shock or other signs of significant heart failure such as rales over the lungs
22. Active or recent (within 1 month prior to study enrollment) participation in another investigational clinical research study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Cardiac MRI infarct size | Day 4
  reduction in infarct size as a percentage of left ventricle size in the per protocol population.

SECONDARY OUTCOMES:
MRI infarct size | Day 4
  Infarct size as percent of area at risk determined with T2-weighted MRI in per protocol population
Myocardial necrosis | 24 Hours
  CK-MB release through 24 hours as area under the curve
NYHA/AHA Cardiac Functional Class | Day 30
  used to describe stages of Heart Failure ( Class I, II, III and IV)
Major Adverse Cardiac Events (MACE) | Month 12
  MACE: Death, MI, re-hospitalization
Angiographic outcomes | Day 1
  TIMI flow grade, TIMI myocardial perfusion grade
ST-segment resolution | Day 1
  ST-segment resolution as a function of time

CONTACTS AND LOCATIONS:
Overall Officials: Goran K Olivecrona, MD, Principal Investigator — Department of Cardiology, Lund University Hospital; David Erlinge, MD, PhD, Principal Investigator — Department of Cardiology, Lund University Hospital
Locations (1):
- Department of Cardiology, Lund University Hospital, Lund, Sweden

REFERENCES:
- [Derived] Erlinge D, Gotberg M, Noc M, Lang I, Holzer M, Clemmensen P, Jensen U, Metzler B, James S, Botker HE, Omerovic E, Koul S, Engblom H, Carlsson M, Arheden H, Ostlund O, Wallentin L, Klos B, Harnek J, Olivecrona GK. Therapeutic hypothermia for the treatment of acute myocardial infarction-combined analysis of the RAPID MI-ICE and the CHILL-MI trials. Ther Hypothermia Temp Manag. 2015 Jun;5(2):77-84. doi: 10.1089/ther.2015.0009. Epub 2015 May 18. PMID 25985169
- [Derived] Erlinge D, Gotberg M, Grines C, Dixon S, Baran K, Kandzari D, Olivecrona GK. A pooled analysis of the effect of endovascular cooling on infarct size in patients with ST-elevation myocardial infarction. EuroIntervention. 2013 Apr 22;8(12):1435-40. doi: 10.4244/EIJV8I12A217. PMID 23164721
- [Derived] Gotberg M, Olivecrona GK, Koul S, Carlsson M, Engblom H, Ugander M, van der Pals J, Algotsson L, Arheden H, Erlinge D. A pilot study of rapid cooling by cold saline and endovascular cooling before reperfusion in patients with ST-elevation myocardial infarction. Circ Cardiovasc Interv. 2010 Oct;3(5):400-7. doi: 10.1161/CIRCINTERVENTIONS.110.957902. Epub 2010 Aug 24. PMID 20736446